CLINICAL TRIAL: NCT04309461
Title: Implementing the Make Better Choices 2 mHealth Energy Balance Intervention for Rural Appalachians
Brief Title: Make Better Choices 2 for Rural Appalachians
Acronym: MBC2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nancy Schoenberg (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Nancy Schoenberg, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 47917; R01HL152714 (NIH)
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Health Behavior
Keywords: app; coaching; Appalachian
MeSH Terms: conditions — Health Behavior; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Management Group (Active Comparator): The Stress Management Program will utilize a smart phone app, accelerometers, telephone coaching, and behavioral incentives to target stress, relaxation, and sleep. Participants will wear accelerometers, log hours slept, enter real-time information about their relaxation exercises and stress, and monitor 3 goal thermometers (sleep, relaxation, stress) to meet behavioral targets. The Stress Management Program, including the use of the app and assessments, is identical to the Adapted MBC2 program, with the exception of the content.
  Interventions: Behavioral: Stress Management Control
- Adapted MBC2 Group (Experimental): The Adapted MBC2 Program will utilize a smart phone app, accelerometers, telephone coaching, and behavioral incentives to target fruit and vegetable intake, dietary fat intake, physical activity, and high sedentary leisure screen time. Participants will wear accelerometers, log hours slept, enter real-time information about their relaxation exercises and stress, and monitor goal thermometers to meet targets.
  Interventions: Behavioral: Adapted MBC2 Program

INTERVENTIONS:
Behavioral: Stress Management Control — The Stress Management Program will utilize a smart phone app, accelerometers, telephone coaching, and behavioral incentives to target stress, relaxation, and sleep. Participants will wear accelerometers, log hours slept, enter real-time information about their relaxation exercises and stress, and monitor 3 goal thermometers (sleep, relaxation, stress) to meet behavioral targets. The Stress Management Program, including the use of the app and assessments, is identical to the Adapted MBC2 program, with the exception of the content.
  Arms: Stress Management Group
Behavioral: Adapted MBC2 Program — The Adapted MBC2 Program will utilize a smart phone app, accelerometers, telephone coaching, and behavioral incentives to target fruit and vegetable intake, dietary fat intake, physical activity, and high sedentary leisure screen time. Participants will wear accelerometers, log hours slept, enter real-time information about their relaxation exercises and stress, and monitor goal thermometers to meet targets.
  Arms: Adapted MBC2 Group

SUMMARY:
The program consists of four interconnected components: (1) app, (2) accelerometer, (3) health coaching, and (4) behavioral incentives to increase food and vegetable intake, reduce saturated fat intake, increase physical activity, and decrease sedentary screen time among adults Appalachia Kentuckians.

DETAILED DESCRIPTION:
Rural Appalachians suffer among the worst health profiles in the US including elevated rates of cardiovascular disease. Although a healthy diet and active lifestyle can reduce mortality and morbidity, only 12% of rural Appalachian Kentuckians consume the recommended daily intake for fruits and vegetables and nearly 35% indicate no physical activity. Personal technology is increasingly common in rural Appalachia, presenting a new opportunity to prevent and manage chronic disease. Most (68%) Appalachian Kentuckians have smart phones and reliable internet access (78%). We propose the first (to our knowledge) adapted evidence-based, multicomponent mHealth (mobile health) intervention program among rural Appalachians. The Make Better Choices 2 (MBC2) intervention has produced significant and sustained improvements in diet and physical activity, using personalized health coaching, an app, accelerometer, and financial incentives. Because of sparse local resources, rural Appalachian residents could greatly benefit from access to appropriate virtual resources through health coaching and mHealth.

In this study, 350 participants will be randomized to receive either the adapted MBC2 or a stress management program. The primary outcome, diet and activity improvement, is a composite change score relative to baseline scores for fruit and vegetable (F/V) intake, fat, physical activity, and sedentary leisure screen time.

Adapted MBC2 intervention content:

The program consists of four interconnected components: (1) app, (2) accelerometer, (3) health coaching, and (4) behavioral incentives. These components encompass behavioral and implementation principles-effectiveness, scalability, and synergy and correspond to the Goal Systems Theory, enhanced by sociocultural and environmental considerations.

1. App: As demonstrated in recent research, increasing personal technology use among rural populations provides a new opportunity for health equity. Apps and accelerometers enable connectivity, accountability, and personalization between participants and their coaches. This app includes a decision support system and display that helps participants monitor fruit & vegetable (F/V) intake, moderate-vigorous physical activity, and sedentary screen time relative to their daily target. This daily diet and activity data entry is a core component of the MBC2 intervention rather than an outcome or assessment. The app also transmits this information to a web-based dashboard accessed by coaches, who use it to tailor telephone counseling.

   During the in-person training, participants will be given materials to help in portion size estimation, plus reminders that entries are time and date-stamped to encourage prompt entry. The app involves automatic wireless data uploading, which enables detection of entry error or non-adherence to protocols. Additional procedures to support adherence to personal goals include: a) visual thermometers to provide feedback about intake and expenditure relative to targets; b) ability to access smart phone diet and activity databases to support decision-making about diet and activity choices; c) visual feedback about goal progress throughout the day to guide self-regulation; and d) use of stepped goals to facilitate incremental attainment of targets. Diet and activity data to assess intervention effectiveness will additionally be collected at the assessment periods via REDCap (baseline and months 3 and 9).
2. Accelerometer: Activity monitors also enhance accountability. Our prior work shows that Appalachian residents have high levels of adherence and satisfaction with accelerometers. For the proposed study, participants will be given a gold standard accelerometer, the triaxial Actigraph GT9X. They will wear it on the non-dominant wrist daily during the intervention. The accelerometer collects data on three axes at a 100 Hz sampling rate, which will be sent via API (application program interface) to display minutes of MVPA (moderate-to-vigorous physical activity) on the study smart phone application as feedback to the participant.
3. Telephone coaching has demonstrated scalability (particularly in more isolated rural locations), effectiveness, and greater reach than in-person counseling. In addition to these benefits, during preparatory focus groups, Appalachians indicated that they prefer telephone coaching over group meetings (due to lack of privacy, time-consuming trips) or home visits (too intrusive). Despite these benefits, telephone coaching is associated with more modest behavioral changes that can undermine longer-term behavior change.
4. Behavioral incentives: An incentive is provided weekly to participants in both conditions if their behavioral average meets goal criterion for the correct use of the app (for data collection) and adherence to behavioral targets (F/V consumption, physical activity and sedentary activity or stress management).

ELIGIBILITY:
Inclusion Criteria:

* adults residing in Appalachian Kentucky
* willingness to use smart phone to record and modify diet and activity
* willingness to wear an accelerometer
* consume <4.5 cups fruit/vegetables daily
* consume >8% daily calories from fat
* engage in <150 minutes of moderate-intensity physical activity weekly
* spend >90 minutes daily on non-work, non-education-related sedentary recreational use of screen time.

Exclusion Criteria:

* unstable medical conditions
* cognitive impairment
* hospitalization for psychiatric disorder within the last 5 years
* active suicidal ideation
* substance use disorder other than nicotine dependence
* at risk for adverse cardiovascular events with moderate-intensity activity
* taking weight loss medication
* trying to get pregnant, pregnant or lactating
* active eating disorders
* using mobility assistive devices
* inability to read study materials

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in diet and activity | 9 months (at baseline, 3 months and 9 months)
  A single composite MBC (Make Better Choices) score of four behaviors (fruit and vegetable intake, fat intake, physical activity, and sedentary screen time) will be used to assess change across multiple diet and activity behaviors. Fruit and vegetable intake, saturated fat intake, and screen time will be measured from smart phone data. Time spent in moderate/vigorous physical activity will be transmitted from the accelerometer to the app. The MBC score, expressing each participant's overall change across the multiple diet and activity behaviors relative to baseline is calculated as the mean of four behavioral individual Z scores at each time point. Scores have an unlimited range; higher values represent greater healthy lifestyle improvement relative to the overall baseline distribution.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life | 9 months (at baseline, 3 months and 9 months)
  The SF-36 (Short Form-36) Health Outcomes Survey will be used to assess patient-reported health. The SF-36 consists of 8 scaled scores, which are weighted sums of the questions in their section. Scores range from 0-100; lower scores indicate more disability.
Change in Blood Pressure | 9 months (at baseline, 3 months and 9 months)
  Sitting total (diastolic and systolic) pressure will be measured according to the CARDIA protocol.
Change in Weight | 9 months (at baseline, 3 months and 9 months)
  Weight will be measured without shoes, wearing a standard hospital gown on a calibrated beam balance scale.
Change in Height | 9 months (at baseline, 3 months and 9 months)
  Height will be measured using a stadiometer.
Change in Body Mass Index (BMI) | 9 months (at baseline, 3 months and 9 months)
  Body Mass Index (BMI) will be calculated as weight in pounds/ (height in inches)^2) x 704.5 and the difference will be calculated.
Change in Waist Circumference | 9 months (at baseline, 3 months and 9 months)
  Waist circumference will be assessed twice during expiration, taking the average for analyses, by positioning an anthropometric tape midway between the palpated iliac crest and the palpated lowest rib margin in the mid-axillary lines.

OTHER OUTCOMES:
Change in total cholesterol | 9 months (at baseline, 3 months and 9 months)
  A12 hour fasting blood sample will be collected for a lipid panel and the change in total cholesterol will be calculated.
Change in triglycerides | 9 months (at baseline, 3 months and 9 months)
  A12 hour fasting blood sample will be collected for a lipid panel and the change in triglycerides will be calculated.
Change in HDL-C | 9 months (at baseline, 3 months and 9 months)
  A12 hour fasting blood sample will be collected for a lipid panel and the change in HDL-C will be calculated.
Change in LDL-C | 9 months (at baseline, 3 months and 9 months)
  A12 hour fasting blood sample will be collected for a lipid panel and the change in LDL-C will be calculated.
Change in plasma glucose | 9 months (at baseline, 3 months and 9 months)
  A12 hour fasting blood sample will be collected and the change in glucose will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Schoenberg, PhD, Principal Investigator — University of Kentucky
Locations (1):
- MBC2 Field Office University of Kentucky, Benham, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vos SC, Adatorwovor R, Roberts MK, Sherman DL, Bonds D, Dunfee MN, Spring B, Schoenberg NE. Community engagement through social media: A promising low-cost strategy for rural recruitment? J Rural Health. 2024 Jun;40(3):467-475. doi: 10.1111/jrh.12809. Epub 2023 Nov 20. PMID 37985592
- [Derived] Nichols CE, Davis J. The Women Farmer Stress Inventory: Examining women farmer stress in the United States Corn Belt. J Rural Health. 2024 Jun;40(3):457-466. doi: 10.1111/jrh.12808. Epub 2023 Nov 14. PMID 37962323
- [Derived] Schoenberg NE, Sherman D, Pfammatter AF, Roberts MK, Chih MY, Vos SC, Spring B. Adaptation and study protocol of the evidence-based Make Better Choices (MBC2) multiple diet and activity change intervention for a rural Appalachian population. BMC Public Health. 2022 Nov 8;22(1):2043. doi: 10.1186/s12889-022-14475-0. PMID 36348358